CLINICAL TRIAL: NCT06090344
Title: Designing Multimedia Patient Education Materials for Adolescent Idiopathic Scoliosis: a Feasibility Randomised Controlled Trial of Patient Education Videos
Brief Title: Designing Multimedia Patient Education for Adolescent Idiopathic Scoliosis
Acronym: PEMAIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Responsible Party: Principal Investigator, Garett Van Oirschot, Principal Investigator, University College Dublin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LS-23-15-VanOirschot-Doherty
Record Dates: First submitted 2023-10-09; First posted 2023-10-19 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Adolescent Idiopathic Scoliosis; Patient Engagement
Keywords: Scoliosis; Multimedia; Patient Education; Health Education; Adolescent Idiopathic Scoliosis
MeSH Terms: conditions — Patient Participation; Scoliosis; Health Education

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual care (No Intervention): Usual care from healthcare providers
- Traditional video format (Experimental): Multimedia videos formatted as traditionally found online
  Interventions: Other: Traditional video format
- Evidence-informed video format (Experimental): Multimedia videos formatted as per evidence advice
  Interventions: Other: Evidence-informed video format

INTERVENTIONS:
Other: Traditional video format — 6 x 3 minute videos designed in the same format as traditionally found on the internet
  Arms: Traditional video format
Other: Evidence-informed video format — 6 x 3 minute videos designed in the format recommended by advice in the literature
  Arms: Evidence-informed video format

SUMMARY:
The goal of this triple-masked three-armed feasibility randomised controlled trial is to compare patient education materials for participants with adolescent idiopathic scoliosis. The main question it aims to answer are:

* Are educational videos superior to usual care?
* Are educational videos formatted in line with literature advice on multimedia design superior to videos formatted as traditionally found on scoliosis advisory websites Participants in the video groups will be asked to do view six educational videos and respond to a quiz. Researchers will compare the informed video group and traditional video group to usual care to see if there are differences in engagement, quality of life, physical activity and health-related anxiety.

DETAILED DESCRIPTION:
Multimedia patient education materials are increasingly used in healthcare. This triple-masked three-armed feasibility randomised controlled trial will examine participants aged 10-18 with radiographically confirmed adolescent idiopathic scoliosis and their response to usual care or to receive multimedia educational videos with or without evidence-informed design principles. Primary outcomes will be patient knowledge measured by online quiz and engagement measured by YouTube analytics. Participants will be masked in the two video intervention arms, as will the therapist sending the educational videos. The results will outline the number of participants recruited and randomised, the number analysed post-intervention and at week eight, and the outcomes for baseline, post-intervention and week 8, which will include the effect size and level of precision. Adverse events will also be reported.

This feasibility randomised controlled trial will offer insight into the effectiveness of implementing advice from the literature in designing multimedia patient education materials for a population with adolescent idiopathic scoliosis.

ELIGIBILITY:
Inclusion Criteria:

* aged 10-18 years
* parent/guardian consent for those under 18 years of age
* adolescent Idiopathic Scoliosis (AIS) as confirmed by Cobb angle ≥10deg on plain film radiographs
* able to watch and listen to online educational materials as well as read and complete online surveys

Exclusion Criteria:

- scoliosis due to non-AIS conditions

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2024-01-30 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Number recruited, rejected, randomised, dropped off, completed | Week 0,1,2,3,4,5,6,7,8
  Number of participants enrolled at each stage of recruitment, rejection, randomisation, during study, and upon completion
Dropout reasons | Week 1,2,3,4,5,6,7,8
  Participant reasons for dropping out (if provided)
Outcomes completed | Week 1,2,3,4,5,6,7,8
  Percentage of outcomes completed
Satisfaction with study procedures | Week 8
  Patient response to tailored question about satisfaction with intervention & study process. Question will read "How satisfied were you with the study process?" and participants will score on a 5-point scale with 1 being Very Unsatisfied and 5 being Very Satisfied
Number and type of adverse events | Week 2,3,4,5,6,7,8
  Adverse events

SECONDARY OUTCOMES:
Scoliosis Research Society 22-revised | Week 0, 8
  Scoliosis Research Society 22-item revised questionnaire of health-related quality of life. The SRS-22r measures quality of life across 5 domains - Function (5 questions), Pain (5 questions) Self-Image (5 questions), Mental Health (5 questions), Satisfaction/Dissatisfaction (2 questions). The maximum score in each domain is 5 and minimum score is 1, with higher scores representing greater patient quality of life.
YouTube Average Watch Duration | Week 1,2,3,4,5,6
  Duration of video view
Knowledge Translation | Week 1,2,3,4,5,6
  5-item multiple choice quiz immediately after video watching
Knowledge Retention | Week 8
  40-item multiple choice quiz after 8 weeks
YouTube Watch Percentage | Week 1,2,3,4,5,6,7,8
  Watch time / Total time
YouTube Behavioural Engagement | Week 1,2,3,4,5,6,7,8
  Percent of time on specific segments
YouTube Time to Complete | Week 1,2,3,4,5,6,7,8
  Time relative to completion
YouTube Visits | Week 1,2,3,4,5,6,7,8
  Number of views for the video
YouTube Affective Engagement | Week 1,2,3,4,5,6
  Selecting thumbs up (like) or down (dislike) using like buttons
European Quality of Life 5-Dimension Youth Version | Week 0, 8
  The EQ-5D-Y descriptive system comprises the following five dimensions: mobility, looking after myself, doing usual activities, having pain or discomfort and feeling worried, sad or unhappy. Each dimension has 3 levels: no problems, some problems and a lot of problems. A higher score indicates higher quality of health.
Physical Activity Questionnaire - older Children | Week 0, 8
  Physical Activity Questionnaire for older Children is a a seven-day recall self-administered questionnaire to evaluate moderately to vigorous physical activity in child. A higher score indicates a higher level of physical activity.
State Trait Anxiety Index (Children) | Week 0, 8
  State Trait Anxiety Index for Children is a psychological inventory consisting of 40 self-report items on a 4-point Likert scale. The STAI measures two types of anxiety - state anxiety and trait anxiety. Higher scores are positively correlated with higher levels of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Cailbhe Doherty, PhD, BSc, Study Chair — University College Dublin
Locations (1):
- University College Dublin, Belfield, Dublin 4, Ireland

IPD SHARING:
Plan to Share IPD: Yes
All anonymised data will be available for viewing on OSF
Supporting Information: Study Protocol, SAP
Time Frame: Available from 2025 when data is expected to be compiled and written up and submitted for publication
Access Criteria: All those with the Open Science Framework link will be able to access the anonymised patient data on the project's Open Science Framework page
URL: https://osf.io/5qmf4/

REFERENCES:
- [Derived] Van Oirschot G, Doherty C. Designing multimedia patient education materials for adolescent idiopathic scoliosis: A protocol for a feasibility randomized controlled trial of patient education videos. PLoS One. 2024 May 23;19(5):e0297394. doi: 10.1371/journal.pone.0297394. eCollection 2024. PMID 38781168

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-09): https://cdn.clinicaltrials.gov/large-docs/44/NCT06090344/Prot_SAP_000.pdf